CLINICAL TRIAL: NCT00511173
Title: Warfarin Dosing: Pharmacogenetic Algorithm Compared to Pharmacist's Dosing
Brief Title: Comparison of Warfarin Dosing Using Decision Model Versus Pharmacogenetic Algorithm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-14171
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Atrial Fibrillation; Pulmonary Embolism; Deep Vein Thrombosis
Keywords: mechanical valve
MeSH Terms: conditions — Atrial Fibrillation; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinician dosing of warfarin (Experimental): Warfarin dose based on clinician dosing without the use of warfarin pharmacogenetics
  Interventions: Genetic: Warfarin Dose based on pharmacogenetics

INTERVENTIONS:
Genetic: Warfarin Dose based on pharmacogenetics — Warfarin dose adjustment will be based on the standard clinician dosing compared to the use of the pharmacogenetic base algorithm

SUMMARY:
This is a prospective comparison of clinician dosing and a pharmacogenetic algorithm in diagnosed patients requiring warfarin therapy.

DETAILED DESCRIPTION:
Diagnosed patients with atrial fibrillation, pulmonary embolism, or deep venous thrombosis requiring warfarin therapy will be consented and a tube of blood for DNA analysis will be drawn. The clinician dosing group will not be eligible to obtain the pharmacogenetic results and the algorithm group will have their warfarin pharmacogenetic SNPs performed and integrated into the algorithm and the warfarin dose will be calculated. Outcomes of patients receiving both methods will be gathered and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed patients with atrial fibrillation, deep venous thrombosis, or pulmonary embolism requiring warfarin therapy

Exclusion Criteria:

* Patients with atrial fibrillation, deep venous thrombosis, or pullmonary embolism requiring warfarin therapy who do not consent to participate

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. Destache, Pharm. D., Principal Investigator — Creighton University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from the warfarin clinic at the Creighton Cardiac Center from 7/06-6/07.
Groups:
- Pharmacist Dosing: Warfarin dose based on pharmacist dosing
Period: Overall Study
Arm/Group | Pharmacist Dosing
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacist Dosing
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (12.3)
Age Continuous [Median (Full Range); unit: years] — Age greater than 40 years
  years | 70 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 56
Region of Enrollment [Number; unit: participants]
  United States | 102
Baseline INR [Mean (Standard Deviation); unit: ratio] | 2.6 (.4)
warfarin dose [Mean (Standard Deviation); unit: mg/wk] | 35.4 (16.4)

OUTCOME MEASURES:

1. Primary Outcome: In Patients Receiving Warfarin, a Pharmacogenetic Algorithm Dose Was Compared to Clinician Dosing (mg/wk).
Description: Warfarin pharmacogenetic algorithm dosing (mg/wk) was compared to clinician warfarin dosing (mg/wk).
Time Frame: six months
Population: power analysis based on data from Sconce, et al.
Measure: Mean (Standard Deviation); unit: mg/wk
Groups:
- Algorithm Dosing: Warfarin dose based on algorithm by Sconce, et al.
- Pharmacist Dosing: Warfarin dose based on clinician dosing
Arm/Group | Algorithm Dosing | Pharmacist Dosing
Number analyzed (Participants) | 102 | 102
mg/wk | 46.9 (7.5) | 35.4 (16.4)
Statistical Analysis 1: Comparison: Algorithm Dosing vs Pharmacist Dosing; Null hypothesis: there is no difference in warfarin dose (mg/wk) between pharmacist dosing and algorithm dosing. In order to gather all SNP groups, the power analysis resulted in > 100 patients enrolled into each group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 10, Standard Deviation 4.5

ADVERSE EVENTS:
Arm/Group | Pharmacist Dosing
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes